CLINICAL TRIAL: NCT03776110
Title: Phase I, Single-center, Multiple Dose, Dose Escalation Study (Within Dose-group Randomised, Double-blind, Placebo-controlled, 2-way Cross-over) to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GRT9906 Prolonged Release Tablets in Healthy Male and Female Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GRT9906 Prolonged Release Tablets After Dose Escalation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP9906-07
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Pharmacokinetics
Keywords: Dose escalation

STUDY DESIGN:
Intervention Model Description: Single center, multiple dose, dose escalation (within dose-group randomized, double-blind, placebo-controlled, 2-way cross-over)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GRT9906 80-mg dose group (Experimental): In one period, 80 mg GRT9906 (2 GRT9906 PR tablets) were administered twice daily at 12 hours apart with non-carbonated water. A total of 7 doses were administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4.
  In the second period, a total of 7 doses of placebo (2 tablets per dose) was administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4.
  Interventions: Drug: GRT9906 PR tablet; Drug: Placebo
- GRT9906 120-mg dose group (Experimental): In one period, 120 mg GRT9906 (3 GRT9906 PR tablets) were administered twice daily at 12 hours apart with non-carbonated water. A total of 7 doses were administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4. A 'titration dose' of 80 mg was administered on the day before Day T. The dose administration on Day T was also performed twice daily with 12 hours apart and with non-carbonated water.
  In the other period, a total of 7 doses of placebo (3 tablets per dose) was administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4.
  Interventions: Drug: GRT9906 PR tablet; Drug: Placebo
- GRT9906 160-mg dose group (Experimental): In one period, 160 mg GRT9906 (4 GRT9906 PR tablets) were administered twice daily at 12 hours apart with non-carbonated water. A total of 7 doses were administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4. A 'titration dose' of 80 mg was administered on Day T. The dose administration on Day T was also performed twice daily with 12 hours apart and with non-carbonated water.
  In the other period, a total of 7 doses of placebo (4 tablets per dose) was administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4.
  Interventions: Drug: GRT9906 PR tablet; Drug: Placebo
- GRT9906 200-mg dose group (Experimental): In one period, 200 mg GRT9906 (5 GRT9906 PR tablets) were administered twice daily at 12 hours apart with non-carbonated water. A total of 7 doses were administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4. A 'titration dose' of 120 mg was administered on Day T. The dose administration on Day T was performed twice daily with 12 hours apart and with non-carbonated water.
  In the other period, a total of 7 doses of placebo (5 tablets per dose) was administered with the first administration in the morning of Day M1 and the last administration in the morning of Day M4.
  Interventions: Drug: GRT9906 PR tablet; Drug: Placebo

INTERVENTIONS:
Drug: GRT9906 PR tablet — 40 mg GRT9906 PR tablet oral (minimal release of 80 percent after 480 minutes)
Drug: Placebo — Placebo tablet matching 40 mg GRT9906 PR tablet

SUMMARY:
The safety and tolerability of multiple oral administrations of GRT9906 at different doses was investigated in this clinical study. The prolonged-release tablets slowly release the active compound in the intestine. In addition, absorption into the body, distribution, metabolization and excretion of GRT9906 was characterized. Pharmacological effects of GRT9906 in healthy participants was assessed using pupillometry (diameter and reactions of the pupil) and a Cold Pressor Test where pain is measured while hands are placed in icy water for two minutes.

DETAILED DESCRIPTION:
The primary objective of the study was to investigate the safety and tolerability of escalating doses of GRT9906 after multiple oral dose administration of prolonged-release (PR) tablets to healthy male and female participants

Secondary objectives were:

* To evaluate the pharmacokinetics (serum and urine) of escalating doses of GRT9906 after multiple oral dose administration of PR tablets and
* To assess the pharmacodynamic effects of escalating doses of GRT9906 by means of pupillometry and Cold Pressor Test after multiple oral dose administration of PR tablets.

The doses of GRT9906 in this study were 80, 120, 160, and 200 milligrams (mg) twice daily in dose groups 1-4.

Participants were screened within 28 days prior to the first dosing. Treatment periods consisted of 5.6 (first dose group) or 6.6 (second and subsequent dose groups) days:

* Day 0 was the day prior to first dosing
* Day T was the titration day (day before Day M1; not applicable for the 80 mg dose group)
* Days M1 to M4 were the days with repeated dosing
* Days F1 and F2 were the follow-up days (24 hours and 48 hours after the last drug administration)
* A final examination was performed within 4 to 14 days after last dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian participants aged 45-70 years;
* Body Mass Index (BMI) between 18 and 30 kilograms per square meter (extremes included);
* Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), electroencephalogram (EEG), vital signs and clinical laboratory parameters (haematology, sedimentation rate, clotting, clinical chemistry, urinalysis and virus serology). Minor deviations of laboratory values and ECG parameters from the normal range may be accepted, if judged by the investigator to have no clinical relevance and if not considered to interfere with the study objectives;
* Adequate contraception. For females of childbearing potential (i.e., all females except surgically sterilized or at least 2 years postmenopausal) this was defined as follows: any form of hormonal contraception or intra-uterine device had to be used, at least from 4 weeks prior to the first dosing up to 4 weeks after the last dosing and an additional barrier contraception (condom or diaphragm) had to be used from 2 weeks prior to the first dosing up to 4 weeks after the last dosing;
* Participants must give written informed consent to participate within this study;
* Negative human immunodeficiency virus-1/2-antibodies, surface antigen of the hepatitis B virus (HBs-antigen), hepatitis B core (HBc)-antibodies, hepatitis C virus (HCV)-antibodies determined at screening examination;
* Negative drug abuse screening test determined at screening examination and prior to first dose administration in each period (the test will include screening for amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids and opiates);
* Negative blood beta-human chorionic gonadotropin (beta-HCG) test for females of childbearing potential determined at screening examination and prior to first dose administration in each period (the test is not necessary in females who are in post-menopausal state for at least 2 years or in females with status after surgical sterilisation).

Exclusion Criteria:

* Pulse rate below 50 or above 100 beats per minute. The measurement must be performed in supine position after a resting period of at least 5 minutes
* Systolic blood pressure below 100 or above 160 millimeters Mercury (mmHg), diastolic blood pressure below 50 or above 100 mmHg. The measurement must be performed in supine position after a resting period of at least 5 minutes;
* Participants with history or presence of diseases or functional disorders of the central nervous system, endocrinological system, gastrointestinal tract, connective tissue, hepatobiliary system, renal system, respiratory system or cardiovascular system or other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs;
* Marked repolarisation abnormality (e.g., suspicious or definite congenital long QT syndrome) or co-medication that is known to influence cardiac repolarisation substantially;
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness); abnormal, clinically relevant EEG findings at screening;
* History of orthostatic hypotension;
* Bronchial asthma;
* Definite or suspected history of drug allergy or hypersensitivity;
* History of Raynaud´s disease or phenomenon;
* Malignancy;
* Participation in another clinical study within the last 3 month prior to the start of this study (exception: characterisation of metaboliser status);
* Blood donation (above 100 milliliters [mL]) or comparable blood losses within three month prior to the start of this study;
* Excessive consumption of food or beverages containing caffeine or other xanthines (more than 1000 mL coffee or equivalent per day) within 2 weeks before administration of the investigational products or during the study;
* Drinking of alcohol containing beverages within 48 hours before administration of the investigational products or during the study;
* Evidence of alcohol, medication or drug abuse;
* Smoking of more than 3 cigarettes per day. Smokers who are not able to abstain from smoking for 24 hours prior to the administration of any cold pressor test, and during the period of hospitalisation must be excluded;
* Intake of drugs that are substrates to cytochrome P2D6 (CYP2D6) isoenzyme within the last 4 weeks prior to the start of this study. Intake of more than 1000 mg paracetamol within 3 days prior to administration of the investigational products. Use of any other medication within 4 weeks prior to the start of the study (self-medication or prescription), if not on a stable basis;
* Neurotic personality, psychiatric illness or suicide risk;
* Known or suspected of not being able to comply with the study protocol or of not being able to communicate meaningfully with the investigator and staff;
* Participants who in the opinion of the investigator should not participate in the study;
* Not able to perform the Cold Pressor Test reproducibly, i.e., the difference in the area under the pain-time curves (AUC) is above 20 percent during the 2 tests performed to evaluate the reproducibility at screening;
* Not able to perform the Vienna Test System (Determination Test, Visual Pursuit Test, Tachistoscopic Traffic Test Mannheim for Screen or equivalent subtests);
* Pregnant or breastfeeding women.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-09-15 (Actual); Primary Completion 2005-03-23 (Actual); Study Completion 2005-03-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events | From Day M1/T (first dose) to Day F2 (5.6 or 6.6 days after first dose)
  Treatment emergent adverse events were collected from first dose of investigational medicinal product (IMP) throughout each treatment period up to and including the 48-hour assessment at the second follow-up day (F2) which was performed after 5.6 days (first dose group) or 6.6 days (second and subsequent dose groups).

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUC0-inf) of GRT9906 after first dose | On Day M1/T (pre-dose and from 0.5 to 12 hours post-dose [11 timepoints in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. AUC0-inf values were calculated by dose group.
Maximum plasma concentration (Cmax) of GRT9906 after first dose | On Day M1/T (pre-dose and from 0.5 to 12 hours post-dose [11 timepoints in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Mean Cmax values were calculated by dose group.
Terminal half life (t half) of GRT9906 after first dose | On Day M1/T (pre-dose and from 0.5 to 12 hours post-dose [11 timepoints in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Mean t half values were calculated by dose group.
Time to maximum serum concentration (tmax) of GRT9906 after first dose | On Day M1/T (pre-dose and from 0.5 to 12 hours post-dose [11 timepoints in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Tmax values were calculated by dose group based on serum concentration data and actual sampling times.
Apparent volume of distribution during the terminal phase (Vz/f) of GRT9906 after first dose | On Day M1/T (pre-dose and from 0.5 to 12 hours post-dose [11 timepoints in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Vz/f was calculated based taking dose, area under the serum concentration-time curve and lambda z into account.
Apparent volume of distribution during the terminal phase (Vz/f) of GRT9906 at steady state | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Vz/f was calculated based taking the maintenance dose, area under the serum concentration-time curve at steady state (AUCss,τ) and lambda z into account.
Area under the concentration time curve in dosing interval τ at steady-state (AUCss,τ) of GRT9906 after last dose | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. The AUCss,τ was calculated by dose group based on the serum concentration time profile.
Area under the concentration time curve at steady-state (AUCss) of GRT9906 after last dose | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. The AUCss was calculated by dose group based on the serum concentration time profile.
Maximum plasma concentration (Cmax) of GRT9906 after last dose | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Mean Cmax values were calculated by dose group.
Time to maximum plasma concentration (tmax) of GRT9906 after last dose | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Tmax values were calculated by dose group based on serum concentration data and actual sampling times.
Terminal half life (t half) of GRT9906 after last dose | On Day M4 (pre-dose and 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Mean t half values were calculated by dose group.
Minimum and maximum steady state concentrations of GRT9906 (Css,min and Css,max) | On Day M4 (pre-dose and from 0.5 to 48 hours post-dose [15 time points in total])
  Serum concentrations of GRT9906 were determined using validated analytical methods. Steady-state minimum and maximum plasma concentration values were calculated by dose group.
Renal clearance (CL/f) of GRT9906 after first dose | On Day M1/T (0.5 hours pre-dose and from 0-2, 2-6, 6-12 hours post-dose)
  Urine concentrations of GRT9906 were determined using validated analytical methods. CL/f was calculated by dose group. Urine samples were collected 0.5 hours before drug administration, and from 0 to 2 hours, 2 to 6 hours, and 6 to 12 hours thereafter.
Renal clearance (CL/f) of GRT9906 after last dose | On Day M1/T (0.5 hours pre-dose); on Day M4 (from 0-2, 2-6, 6-12, 12-24, 24-36, and 36-48 hours post-dose)
  Urine concentrations of GRT9906 were determined using validated analytical methods. CL/f was calculated by dose group. Samples were collected 0.5 hours before first drug administration and on Days M4 from 0 to 2 hours, 2 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours.
Changes in static and dynamic pupillometry parameters: initial pupil diameter and amplitude | On Days T/M1 and M4 (-1, 1, 2, 3, 4, 6, 8 and 12 hours after morning dose); on Day F1 (i.e., 24 hours after last dosing on Day M4)
  Static and dynamic pupillometry was performed to assess dose-related decreases in pupillary size and the velocity of reaction to a light stimulus. All assessments were conducted in an invariably darkened room. Initial pupil diameter (mm) and amplitude of constriction (mm) were determined.
Changes in static and dynamic pupillometry parameters: latency and constriction time | On Days T/M1 and M4 (-1, 1, 2, 3, 4, 6, 8 and 12 hours after morning dose); on Day F1 (i.e., 24 hours after last dosing on Day M4)
  Static and dynamic pupillometry was performed to assess dose-related decreases in pupillary size and the velocity of reaction to a light stimulus. All assessments were conducted in an invariably darkened room. Onset latency of myosis (milliseconds) and constriction time (milliseconds) were determined.
Changes in the area under the pain-time curve (AUCcpt) using the Cold Pressor Test | On Day M3 (before dosing and 2, 4 and 8 hours after the morning dose)
  The participant's dominant hand is immersed into a 1-3 degrees Celsius circulating water quench for 2 minutes. Pain intensity is documented on a visual analogue scale (from "no pain" to "maximum pain") on a computer screen facing the participant, using the arrow keys on the keyboard. The participant moves the pointer across the line to rate their feelings at the time. The AUCcpt was assessed after IMP administration; changes to baseline (before dosing) were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- FOCUS Clinical Drug Development GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No